CLINICAL TRIAL: NCT02723994
Title: A Phase 2 Study of the JAK1/JAK2 Inhibitor Ruxolitinib With Chemotherapy in Children With De Novo High-Risk CRLF2-Rearranged and/or JAK Pathway-Mutant Acute Lymphoblastic Leukemia
Brief Title: A Phase 2 Study of Ruxolitinib With Chemotherapy in Children With Acute Lymphoblastic Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Collaborators: Children's Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 18424-269; AALL1521 (Other: Children's Oncology Group)
Expanded Access: NCT03147742 (Approved for marketing)
Record Dates: First submitted 2016-03-09; First posted 2016-03-31 (Estimated); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Leukemia
Keywords: B-cell acute lymphoblastic leukemia (ALL); pediatric; multi-agent chemotherapy; JAK inhibitor
MeSH Terms: conditions — Leukemia; Burkitt Lymphoma | interventions — ruxolitinib; asparaginase erwinia chrysanthemi recombinant; Cyclophosphamide; Cytarabine; Dexamethasone; Doxorubicin; Leucovorin; Mercaptopurine; Methotrexate; pegaspargase; Prednisone; Thioguanine; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ruxolitinib in combination with chemotherapy (Experimental)
  Interventions: Drug: Ruxolitinib; Drug: Asparaginase Erwinia Chrysanthemi; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin; Drug: Leucovorin Calcium; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Drug: Prednisone; Drug: Thioguanine; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Ruxolitinib — In Part 1, ruxolitinib will be administered at a protocol-defined starting dose in combination with chemotherapy, with dose escalation and de-escalation following the rolling 6 study design. The established recommended starting dose will be taken forward into Part 2.
  Other Names: INCB018424
Drug: Asparaginase Erwinia Chrysanthemi
Drug: Cyclophosphamide
Drug: Cytarabine
Drug: Dexamethasone
Drug: Doxorubicin
Drug: Leucovorin Calcium
Drug: Mercaptopurine
Drug: Methotrexate
Drug: Pegaspargase
Drug: Prednisone
Drug: Thioguanine
Drug: Vincristine Sulfate

SUMMARY:
This is a nonrandomized study of ruxolitinib in combination with a standard multi-agent chemotherapy regimen for the treatment of B-cell acute lymphoblastic leukemia. Part 1 of the study will optimize the dose of study drug (ruxolitinib) in combination with the chemotherapy regimen. Part 2 will evaluate the efficacy of combination chemotherapy and ruxolitinib at the recommended dose determined in Part 1.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for study when participant is 1 year to 21 years at the time of diagnosis
* Eligible Ages in Canada; 2 years to 21 years
* De novo high-risk (HR) Ph-like B-ALL for which any of following criteria are present at diagnosis:

  * Age ≥ 10 years
  * White blood cell (WBC) ≥ 50 × 10^3/μL
  * CNS3 leukemia at diagnosis
  * Systemic steroid pretreatment without presteroid WBC documentation
* Diagnostic bone marrow or peripheral blood sample must have gene expression profiling and downstream genetic testing performed by submitting diagnostic specimens under the COG AALL08B1 or APEC14B1 biology studies, or AALL1131 or its successor study. Specimens must demonstrate a Ph-like expression profile (ie, LDA-positive) as tested by low density microarray testing at the COG ALL reference laboratory or TriCore laboratory at the University of New Mexico AND must contain 1 of the following genetic lesions: (determined at COG ALL reference laboratories, or equivalent CAP/CLIA-certified laboratories approved by the medical monitor:

  1. CRLF2 rearrangement with confirmed JAK1 or JAK2 mutation (JAK+)
  2. CRLF2 rearrangement without JAK mutation
  3. Other JAK pathway alterations (eg, JAK2 fusions, EPOR fusions, SH2B3 deletions, IL7RA mutations) with or without CRLF2-R, or CRLF2-R with unknown JAK status as determined by a COG ALL Reference Laboratory
* Completed a 4-drug Induction therapy regimen (modified aBFM regimen or equivalent) in Study AALL1131 or its successor study, or as per the institutional standard of care for HR B-ALL and have had end-Induction minimal residual disease (MRD) assessed
* Male and female subjects of reproductive non childbearing potential or willing to take appropriate precautions to avoid pregnancy or fathering a child for the duration of study participation

Exclusion Criteria:

* Receipt of any other cytotoxic chemotherapy before Induction therapy, with exception of hydroxyurea or steroid pretreatment
* Trisomy 21 (Down syndrome)
* BCR-ABL1-rearranged (Ph+) ALL
* Calculated creatinine clearance or radioisotope glomerular filtration rate < 70 mL/min/1.73 m^2
* Alanine aminotransferase ≥ 5 × upper limit of normal (ULN) for age
* Direct bilirubin ≥ 1.5 × ULN (may be assumed if total bilirubin is below ULN)
* History or evidence of cirrhosis
* Platelet count < 75 × 10^3/μL
* Absolute neutrophil count (ANC) < 750/μL
* Positive screen for hepatitis B or C
* Known human immunodeficiency virus infection

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 171 (Actual)
Dates: Start 2016-09-30 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Part 1: Safety/tolerability of ruxolitinib in combination with chemotherapy as measured by adverse events (AEs), vital signs, clinical laboratory tests, and echocardiograms | Part 1: AEs assessed from screening through up to 30 days after the last dose of study drug, expected to be 26 months (females) or 38 months (males)
Part 2: Efficacy of ruxolitinib in combination with chemotherapy as measured by Event-free survival, defined as the percentage of patients alive without relapse, progression, or death at 3 years from study Day 1 | Part 2: assessed at 3 years

SECONDARY OUTCOMES:
Safety and tolerability of the combination treatment for subjects beginning treatment at the recommended dose for Part 2, as assessed by AEs, vital signs, clinical laboratory tests, and echocardiograms | AEs assessed from screening through up to 30 days after the last dose of study treatment, expected to be 26 months (females) or 38 months (males)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Assad, MD, Study Director — Incyte Corporation; Sarah Tasian, MD, Study Chair — Children's Hospital of Philadelphia, Philadelphia, PA
Locations (111):
- United States (103):
  - The Childrens Hospital of Alabama, Birmingham, Alabama
  - Phoenix Children'S Hospital, Phoenix, Arizona
  - Arkansas Childrens Hospital, Little Rock, Arkansas
  - Kaiser Permanente, Fontana, California
  - Loma Linda University Cancer Center, Loma Linda, California
  - Miller Childrens Hospital Pharmacy, Long Beach, California
  - Children'S Hospital Los Angeles, Los Angeles, California
  - Kaiser Foundation Health Plan, Los Angeles, California
  - Southern California Permanente Medical Group, Los Angeles, California
  - Valley Childrens Hospital, Madera, California
  - Choc Children Hospital, Orange, California
  - Lucille Packard Childrens Hospital, Palo Alto, California
  - Kaiser Permanente, San Diego, California
  - Rady Children'S Hospital - San Diego, San Diego, California
  - Ucsf Pediatric Oncology, San Francisco, California
  - Kaiser Permanente Downey, Santa Fe Springs, California
  - Children'S Hospital Colorado, Aurora, Colorado
  - Connecticut Children'S Medical Ctr, Hartford, Connecticut
  - Smilow Cancer Center - Yale, New Haven, Connecticut
  - Alfred I. Dupont Hospital For Children, Wilmington, Delaware
  - Childrens Hospital of Southwest Florida, Fort Myers, Florida
  - Joe Dimaggio Children Hospital, Hollywood, Florida
  - Nemours Childrens Clinic, Jacksonville, Florida
  - University of Florida Health Shands Hospital, Jacksonville, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - Arnold Palmer Hospital For Children, Orlando, Florida
  - Nemours Childrens Clinic, Pensacola, Florida
  - All Childrens Hospital, St. Petersburg, Florida
  - St Josephs Childrens Hospital Tampa, Tampa, Florida
  - Saint Marys Medical Center, West Palm Beach, Florida
  - Egleston Children'S Health, Atlanta, Georgia
  - Kapiolani Medical Center For Women and Children, Honolulu, Hawaii
  - Ann & Robert H. Lurie Children'S Hospital, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital For Children, Indianapolis, Indiana
  - St Vincent Hospital, Indianapolis, Indiana
  - Blank Childrens Hospital, Des Moines, Iowa
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Kosair Childrens Hospital, Louisville, Kentucky
  - Ochsner Clinic, New Orleans, Louisiana
  - Maine Center For Cancer Medicine, Scarborough, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Dana Farber Boston Children'S, Boston, Massachusetts
  - Cs Mott Childrens Hospital, Ann Arbor, Michigan
  - Helen Devos Childrens Hosp, Grand Rapids, Michigan
  - Michigan State University, Lansing, Michigan
  - Children'S Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - The Children'S Mercy Hospital Outpatient, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - Children'S Hospital & Medical Center, Omaha, Nebraska
  - Alliance For Childhood Diseases, Las Vegas, Nevada
  - Children'S Center For Cancer & Blood Dis, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of Nj, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - St Josephs Regional Medical Center, Paterson, New Jersey
  - University of New Mexico Hospital, Albuquerque, New Mexico
  - Albany Medical College, Albany, New York
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Cohen Children'S Medical Center, New Hyde Park, New York
  - Weill Cornell Medical College, New York, New York
  - Nyu Clinical Cancer Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Suny Upstate Medical University, Syracuse, New York
  - New York Medical College, Valhalla, New York
  - University of North Carolina At Chapel Hill, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Akron Children'S Hospital, Akron, Ohio
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies & Children Hosp, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children'S Hospital, Columbus, Ohio
  - Dayton Children'S Hospital, Dayton, Ohio
  - Toledo Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Doernbecher Childrens Hospital, Portland, Oregon
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Children'S Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Childrens Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Hasbro Childrens Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Dell Childrens Medical Center of Central Texas, Austin, Texas
  - Driscoll Children'S Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - El Paso Children'S Hospital Corporation, El Paso, Texas
  - Texas Childrens Hospital, Houston, Texas
  - University of Texas Health Science Cente, San Antonio, Texas
  - Primary Children'S Hospital, Salt Lake City, Utah
  - Children'S Hospital of the, Norfolk, Virginia
  - Seattle Children'S Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center & Children'S Hospital, Spokane, Washington
  - St Vincent Hospital, Green Bay, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (6):
  - Alberta'S Children Hospital, Calgary, Alberta
  - Bc Children'S Hospital, Vancouver, British Columbia
  - The Hospital For Sick Children, Toronto, Ontario
  - Chu Sainte-Justine, Montreal, Quebec
  - McGill University Health Centre/Glen Site/Cedars Cancer Centre, Montreal, Quebec
  - McMaster University Medical Centre, Hamilton
- Puerto Rico (2):
  - University Pediatric Hospital, San Juan, PR
  - San Jorge Childrens Hospital, San Juan